CLINICAL TRIAL: NCT00810108
Title: Pharmacokinetics of Lopinavir Crushed Versus Whole Tablets in Pediatric Patients
Brief Title: Lopinavir/Ritonavir (Kaletra) PK in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: American Association of Colleges of Pharmacy (Other)
Responsible Party: Principal Investigator, Brookie Best, PharmD, MAS, Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10894
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Results first posted 2012-07-06 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-06

CONDITIONS: HIV/AIDS Treatment; HIV Infections
Keywords: HIV/AIDS; pediatrics; resource-limited settings; lopinavir; ritonavir; Kaletra®; antiretroviral treatment; crushed tablets; treatment experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Lopinavir; Ritonavir; lopinavir-ritonavir drug combination; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole Then Crushed Tablets (Experimental): These subjects will take whole lopinavir tablets at Study Visit 1, and crushed tablets at Study Visit 2.
  Interventions: Drug: lopinavir/ritonavir (Kaletra®) tablets
- Crushed Then Whole Tablets (Experimental): These subjects will take crushed tablets at Study Visit 1, and whole tablets at Study Visit 2.
  Interventions: Drug: lopinavir/ritonavir (Kaletra®) tablets

INTERVENTIONS:
Drug: lopinavir/ritonavir (Kaletra®) tablets — The subject will bring their own prescription of lopinavir/ritonavir. The patient will take a witnessed dose of lopinavir/ritonavir with an 6 ounce glass of cool water (if taken whole) or mixed in 4 ounces of Jell-O brand pudding (if crushed).
  Other Names: Kaletra®

SUMMARY:
The objective of this study is to compare the pharmacokinetics of lopinavir tablets administered to pediatric patients as either whole or crushed tablets. The study is a randomized,open-label, crossover study of pediatric subjects already taking lopinavir/ritonavir tablets as part of their clinical care. THe investigators hypothesize that lopinavir exposure in pediatric patients will be lower after taking a dose of the tablet formulation, crushed and mixed with pudding or yogurt, as compared to the exposure after taking a dose with tablets swallowed whole.

DETAILED DESCRIPTION:
By the end of 2005, approximately 2.3 million children worldwide were living with HIV/AIDS.1 At least 660,000 children worldwide have advanced HIV/AIDS and are in dire need of antiretroviral treatment. While many barriers exist to scaling up HIV/AIDS care and treatment globally, access to life-saving treatments for children is increasing. The protease inhibitor, lopinavir/ritonavir (Kaletra®), is recommended as a first-line agent by the World Health Organization and by the US Department of Health and Human Services for the treatment of pediatric patients in resource-limited settings and in the United States.

The prescribing information states that these tablets may not be crushed, broken or chewed, and the manufacturer does not plan to examine the pharmacokinetics of crushed tablets at this time. The company found that the crushed tablets were poorly absorbed in a small pharmacokinetic study in several dogs. While this information has spread through investigators by word-of-mouth, this information has not been published in any forum by the company, and no guidance as to the extent of the decrease in absorption has been provided. However, patients and caregivers are dosing pediatric patients with crushed tablets to overcome some of the limitations of the oral solution. If crushed tablet administration yields significantly lower systemic exposure to lopinavir than whole tablets, then patients using this administration technique will be at higher risk for development of viral resistance and treatment failure. This administration technique must be studied so that providers have evidence to support recommendations about this dose administration strategy.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* Taking lopinavir/ritonavir (Kaletra) tablets at standard pediatric doses for greater than two weeks
* Concomitant medications and/or natural products, including potentially interacting products, have been stable for greater than two weeks and are not expected to change over the course of the study
* Ability to understand study procedures and assent to participate
* Parental or guardian consent
* Aged 6 - 17 years

Exclusion Criteria:

* Acute serious medical illness or infection (in the judgment of the investigator)requiring treatment and/or hospitalization within 14 days prior to study entry
* Pregnancy
* Concomitant medications/natural products that have been started within past two weeks and/or that will be changed over the course of the study.

Ages: 6 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2006-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brookie Best, PharmD, MAS, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - University of California, San Diego - Skaggs School of Pharmacy and School of Medicine, San Diego, California
  - Children's National Medical Center, Washington D.C., District of Columbia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between August 2008 to August 2009 from the Special Immunology Program at Children' National Medical Center in Washington DC.
Period: Overall Study
Arm/Group | Whole Then Crushed Tablets | Crushed Then Whole Tablets
Started | 6 | 7
Completed | 5 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Whole Then Crushed Tablets | Crushed Then Whole Tablets | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 7 | 13
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Median (Full Range); unit: Years] | 12 [10 to 16] | 13 [12 to 16] | 13 [10 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Lopinavir Area Under the Curve (AUC)
Description: Lopinavir Area Under the Plasma Concentration versus Time Curve (AUC)
Time Frame: pre-dose, 1,2,4,6,8, and 12 hours post-dose
Population: All subjects who completed the pharmacokinetic sampling visits with whole tablet administration were analyzed
Measure: Median (Inter-Quartile Range); unit: mg*hr/L
Groups:
- All Subjects Taking Whole Tablets: Lopinavir AUC from all subjects taking the whole tablet
- All Subjects Taking Crushed Tablets: Lopinavir AUC from all subjects taking the crushed tablet
Arm/Group | All Subjects Taking Whole Tablets | All Subjects Taking Crushed Tablets
Number analyzed (Participants) | 12 | 12
mg*hr/L | 144 [101 to 202] | 92 [79 to 103]
Statistical Analysis 1: Comparison: All Subjects Taking Whole Tablets vs All Subjects Taking Crushed Tablets; Lopinavir AUC was compared between whole tablet and crushed tablet administration by using a ratio of crushed/whole AUC; Test type: Non-Inferiority or Equivalence — The geometric mean and 90% confidence interval assessed whether the crushed and whole tablet administration AUCs were equivalent; p < 0.05, t-test, 2 sided; Ratio of Crushed/Whole Tablet AUC = 0.55, 90% CI 2-sided [0.45 to 0.69]

ADVERSE EVENTS:
Groups:
- All Subjects: Data from all subjects combined
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

LIMITATIONS AND CAVEATS:
The AUC of the crushed tablet administration were measured after a single dose only, rather than at steady-state; variable adherence may have impacted results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No